CLINICAL TRIAL: NCT05331391
Title: A Brief Mobile SMART Exercise Support Program to Improve Fatigue in Patients With Advanced Lung Cancer - A Pragmatic Randomized Controlled Trial With Outcome and Process Evaluation
Brief Title: A Mobile SMART Exercise Support Program to Improve Fatigue in Lung Cancer Patients - A RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW21-148
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The Experimental group will receive a brief SMART Exercise individual face-to-face session, and a package of information on lifestyle-integrated exercise and physical activity delivered through instant messaging and telephone calls.
  The Control group will receive a face-to-face individual session on general hygiene (GH) information, and a package of information on GH delivered through instant messaging and telephone calls.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor did not aware of which groups the patients belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief mobile SMART Exercise Support Program (Experimental): Patients will receive a brief SMART Exercise individual session with instant messages and telephone coaching for exercise habit formation and maintenance.
  Interventions: Behavioral: Brief mobile SMART Exercise Support Program
- General Hygiene Information (GHI) (Placebo Comparator): Patients will receive an individual session, instant messages and telephone coaching regarding general hygiene information.
  Interventions: Behavioral: Brief mobile SMART Exercise Support Program

INTERVENTIONS:
Behavioral: Brief mobile SMART Exercise Support Program — Patients will receive 1) a brief SMART Exercise individual face-to-face session; 2) a theory-based instant messaging (WhatsApp/WeChat) and telephone-delivered health coaching on a 2-stage tapering schedule. Stage 1 (week 1 to 6): daily messages and two biweekly phone calls for exercise habit formation. Stage 2 (week 7 to 12): messages twice a week and monthly phone calls for exercise habit maintenance.

SUMMARY:
Lung cancer (LC) is a common cancer in the world. Among all symptoms, Fatigue is considered as the most distressing medical condition of LC. Prior studies revealed that physical activity effectively relieve fatigue and related problems. The current study attempt to explore the effectiveness of SMART Exercise Support Program (SES) with the use of mobile instant messaging application, on reducing symptoms such as fatigue, and improving physical activity level, physical fitness performance, sleep quality and habits, and quality of life in advanced lung cancer (ALC) patients.

DETAILED DESCRIPTION:
Lung cancer (LC) is the most and second most common cancer globally and locally, respectively. Nearly half of LC patients are diagnosed in the advanced stage. Fatigue is perceived to be the most distressing symptom. Physical activity has been proposed as an alternative treatment to relieve fatigue and related problems.

Mobile instant messaging applications (e.g. WhatsApp/WeChat) are popular and inexpensive for interactive messaging. A systematic review showed a majority of messaging interventions were effective in diabetes self-management, weight loss, physical activity (PA), smoking cessation, and medication adherence.

The proposed randomized controlled trial (RCT) aims to examine the effectiveness of SES on relieving fatigue, pain, dyspnea, happiness, anxiety and depression symptoms, physical activity level, physical fitness performance, sleep quality and habits, and quality of life in ALC patients (SES group), compared to the General Hygiene Information (GHI, control) group.

Questionnaires and simple fitness tests will be used at baseline, 6-week, and 24-week assessments. Qualitative feedback will be obtained at the completion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above;
* Diagnosis of Stage III or IV non-small cell lung cancer;
* Edmonton Symptom Assessment System Scale fatigue symptom score ≥4 out of 10
* Self-reported engagement of <150 minutes of moderate intensity PA each week,
* Ambulatory and capable of all self-care activities (European Co-operative Oncology Group (ECOG) Performance Status of ≤2)
* Either undergoing or finished oncology therapy, biological agents and/or support care;
* Mentally, cognitively and physically fit to join the trial as determined by the doctor in-charge and responsible clinical investigators;
* Able to speak and read Chinese;
* Willing to complete the patient-reported outcome questionnaire;
* Completion of the Physical Activity Readiness Questionnaire; and
* Possession of a smartphone with instant messaging functions such as WhatsApp or WeChat.

Exclusion Criteria:

* Those preparing for lung operation;
* Skeletal fragility;
* Serious active infection;
* Inability to walk;
* Previously untreated symptomatic brain metastases;
* Severe respiratory insufficiency;
* Uncontrolled pain; or
* Diagnosed psychiatric illness with or without medication such as major depressive disorder.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue level | Baseline and 6 weeks
  Measured by a 13-item Functional Assessment of Cancer Therapy - Fatigue subscale. The level of fatigue is measured on a five-point Likert scale. The scale range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue.

SECONDARY OUTCOMES:
Change in fatigue level | Baseline and 6 months
  Measured by a 13-item Functional Assessment of Cancer Therapy - Fatigue subscale. The level of fatigue is measured on a five-point Likert scale. The scale range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue.
Change in anxiety symptoms | Baseline, 6 weeks, 6 months
  Measured by a 7-item Generalised Anxiety Disorder Assessment. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 21. The higher scores the greater severity of anxiety symptoms.
Change in depression symptoms | Baseline, 6 weeks, 6 months
  Measured by a 9-item Patient Health Questionaire. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 27. The higher scores the greater severity of depression symptoms.
Change in physical activity level | Baseline, 6 weeks, 6 months
  Measured the days and duration of physical activity level and sitting time in the past 7 days by the International Physical Activity Questionnaire (short version) with 4 questions.
Change in sleep quality | Baseline, 6 weeks, 6 months
  Measured by 7-item Severe Insomnia Index. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 28. The higher scores the greater severity of insomnia.
Change in health-related quality of life | Baseline, 6 weeks, 6 months
  Measured by a 30-item European Organization for Research and Treatment of Cancer and Lung Module. It contains five functioning scales (physical, social, role, cognitive, and emotional functioning), and eight symptom scales (fatigue, nausea/vomiting, pain, dyspnea, sleep disturbances, appetite loss, constipation, and diarrhoea), and financial impact, and overall quality of life. All scale scores are linearly converted to a range from 0 to 100. Higher scores indicate better functioning for the functioning scales and global QOL; for the symptom scales, higher scores indicate higher symptom burden.
Change in happiness level | Baseline, 6 weeks, 6 months
  Measured by 4-item Subjective Happiness Scale with a 7-point Likert scale. Total scores range from 4 to 28. The highest scores reflect greater happiness.
Change in cancer-related symptoms | Baseline, 6 weeks and 6 months
  Measured by 3 items of the Edmonton Symptom Assessment System Scale. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity.
Change in acceptance of illness | Baseline, 6 weeks and 6 months
  Measured by a 5-item subscale of Peace, Equanimity, and Acceptance in the Cancer Experience questionnaire
Change in exercise self-efficacy | Baseline, 6 weeks and 6 months
  Measured by a question with a scale from 0 to 10; "0" indicates no exercise self-efficacy, while "10" indicates highest level of exercise self-efficacy.
Change in social and family support | Baseline, 6 weeks and 6 months
  Measured by 8-item family and friend subscales of multidimensional Scale of Perceived Social Support with a 7-point Likert scale. Each scale ranges from 4 to 28. A higher score equates with higher social support.
Change in grip strength | Baseline, 6 weeks and 6 months
  Measured by a dynamometer
Change in lower limb strength | Baseline, 6 weeks, and 6 months
  Measured by 30-second chair stand test.
Change in balance | Baseline, 6 weeks and 6 months
  Measured by single-leg-stance test
Change in flexibility | Baseline, 6 weeks, and 6 months
  Measured by chair sit and reach test
Change in objective physical activity levels, including duration, frequency and intensity | Baseline, 6 weeks, and 6 months
  Measured by a waist-worn accelerometer
Change in sleep and wake intervals | Baseline, 6 weeks , and 6 months
  Measured by watch-like activity monitor
Change in exercise capacity | Baseline, 6 weeks and 6 months
  Measured by a 6-min walk test

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For those who want the patient data, please contact PI directly by written email.

REFERENCES:
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ho RT, Fong TC. Factor structure of the Chinese version of the Pittsburgh sleep quality index in breast cancer patients. Sleep Med. 2014 May;15(5):565-9. doi: 10.1016/j.sleep.2013.10.019. Epub 2014 Feb 18. PMID 24759325
- [Background] Koller M, Hjermstad MJ, Tomaszewski KA, Tomaszewska IM, Hornslien K, Harle A, Arraras JI, Morag O, Pompili C, Ioannidis G, Georgiou M, Navarra C, Chie WC, Johnson CD, Himpel A, Schulz C, Bohrer T, Janssens A, Kulis D, Bottomley A. An international study to revise the EORTC questionnaire for assessing quality of life in lung cancer patients. Ann Oncol. 2017 Nov 1;28(11):2874-2881. doi: 10.1093/annonc/mdx453. PMID 28945875
- [Background] Chie WC, Yang CH, Hsu C, Yang PC. Quality of life of lung cancer patients: validation of the Taiwan Chinese version of the EORTC QLQ-C30 and QLQ-LC13. Qual Life Res. 2004 Feb;13(1):257-62. doi: 10.1023/B:QURE.0000015295.74812.06. PMID 15058806
- [Background] Nan H, Ni MY, Lee PH, Tam WW, Lam TH, Leung GM, McDowell I. Psychometric evaluation of the Chinese version of the Subjective Happiness Scale: evidence from the Hong Kong FAMILY Cohort. Int J Behav Med. 2014 Aug;21(4):646-52. doi: 10.1007/s12529-014-9389-3. PMID 24515396
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Jones CJ, Rikli RE, Max J, Noffal G. The reliability and validity of a chair sit-and-reach test as a measure of hamstring flexibility in older adults. Res Q Exerc Sport. 1998 Dec;69(4):338-43. doi: 10.1080/02701367.1998.10607708. PMID 9864752
- [Background] Newton R. Review of tests of standing balance abilities. Brain Inj. 1989 Oct-Dec;3(4):335-43. doi: 10.3109/02699058909004558. PMID 2684312
- [Background] Santos-Lozano A, Santin-Medeiros F, Cardon G, Torres-Luque G, Bailon R, Bergmeir C, Ruiz JR, Lucia A, Garatachea N. Actigraph GT3X: validation and determination of physical activity intensity cut points. Int J Sports Med. 2013 Nov;34(11):975-82. doi: 10.1055/s-0033-1337945. Epub 2013 May 22. PMID 23700330
- [Background] Bonomi AG, Westerterp KR. Advances in physical activity monitoring and lifestyle interventions in obesity: a review. Int J Obes (Lond). 2012 Feb;36(2):167-77. doi: 10.1038/ijo.2011.99. Epub 2011 May 17. PMID 21587199
- [Background] Kushida CA, Chang A, Gadkary C, Guilleminault C, Carrillo O, Dement WC. Comparison of actigraphic, polysomnographic, and subjective assessment of sleep parameters in sleep-disordered patients. Sleep Med. 2001 Sep;2(5):389-96. doi: 10.1016/s1389-9457(00)00098-8. PMID 14592388